CLINICAL TRIAL: NCT00823992
Title: A Randomized, Double-blind, Placebo-controlled Study to Assess the Effect of Taspoglutide on Glycemic Control, and Its Safety and Tolerability, in Obese Patients With Type 2 Diabetes Mellitus Inadequately Controlled With Metformin Monotherapy.
Brief Title: A Study of Taspoglutide Versus Placebo for the Treatment of Obese Patients With Type 2 Diabetes Mellitus Inadequately Controlled With Metformin Monotherapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BC22092; 2008-005809-20
Record Dates: First submitted 2009-01-15; First posted 2009-01-16 (Estimated); Last update posted 2016-07-28 (Estimated); Status verified 2016-07

CONDITIONS: Diabetes Mellitus Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — taspoglutide

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- placebo (Placebo Comparator)
  Interventions: Drug: placebo
- taspoglutide (Experimental)
  Interventions: Drug: taspoglutide

INTERVENTIONS:
Drug: placebo — sc once weekly
  Arms: placebo
Drug: taspoglutide — 10mg sc once weekly for 4 weeks, then 20mg sc once weekly
  Arms: taspoglutide

SUMMARY:
This 2 arm study will assess the efficacy, safety and tolerability of taspoglutide compared to placebo in obese patients with type 2 diabetes mellitus inadequately controlled with metformin monotherapy. Patients will be randomized to receive taspoglutide (10mg sc once weekly for 4 weeks followed by 20mg once weekly) or placebo sc, in addition to their prescribed, pre-existing metformin therapy.After the first 24 weeks, patients on placebo will be switched to taspoglutide 20mg once weekly (after 4 weeks on taspoglutide 10mg once weekly) The anticipated time on study treatment is 12 months, and the target sample size is 100-500 individuals.

ELIGIBILITY:
Inclusion Criteria:

* adult patients, 18-75 years of age;
* type 2 diabetes mellitus, receiving metformin at a stable dose of >=1500mg/day for at least 12 weeks;
* HbA1c >=6.5% and <=9.5% at screening;
* BMI >=30 and <=50 kg/m2 at screening;
* stable weight +/-5% for at least 12 weeks prior to screening.

Exclusion Criteria:

* history of type 1 diabetes or acute metabolic diabetic complications such as ketoacidosis or hyperosmolar coma within the past 6 months;
* evidence of clinically significant diabetic complications;
* myocardial infarction, coronary artery bypass surgery, post-transplantation cardiomyopathy or stroke within the past 6 months.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 305 (Actual)
Dates: Start 2009-01; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Absolute change from baseline in HbA1c | 24 weeks

SECONDARY OUTCOMES:
Change from baseline in body weight;% of patients achieving >=5% weight loss | 24 weeks
% of patients achieving target HbA1c <=6.5%, <=7.0%; change from baseline in fasting plasma glucose; change from baseline in lipid profile; relative change in glucose, insulin, C-peptide and glucagon during a meal tolerance test; beta cell function | 24 weeks
Safety:Adverse events,clinical laboratory tests, vital signs,physical examination, ECG, anti-taspoglutide antibodies\n | At planned clinic visits, for 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (69):
- United States (29):
  - Bermuda Dunes, California
  - La Jolla, California
  - Los Angeles, California
  - Mission Viejo, California
  - Brooksville, Florida
  - Miami, Florida
  - St. Petersburg, Florida
  - Atlanta, Georgia
  - Chicago, Illinois
  - Avon, Indiana
  - New Orleans, Louisiana
  - Bangor, Maine
  - Royal Oak, Michigan
  - Picayune, Mississippi
  - Clifton, New Jersey
  - Toms River, New Jersey
  - Albuquerque, New Mexico
  - New York, New York
  - Springfield Gardens, New York
  - Charlotte, North Carolina
  - Shelby, North Carolina
  - Norman, Oklahoma
  - Medford, Oregon
  - Clinton, South Carolina
  - Kingsport, Tennessee
  - Dallas, Texas
  - Houston, Texas
  - Midland, Texas
  - San Antonio, Texas
- Canada (6):
  - Vancouver, British Columbia
  - Sherbrooke, Nova Scotia
  - Etobicoke, Ontario
  - Hamilton, Ontario
  - Oakville, Ontario
  - Toronto, Ontario
- Germany (9):
  - Aschaffenburg
  - Berlin
  - Bochum
  - Dortmund
  - Dresden
  - Falkensee
  - Mainz
  - Münster
  - Neuwied
- Italy (4):
  - Ancona
  - Ravenna
  - Roma
  - Siena
- Bitola, North Macedonia
- Poland (3):
  - Gniewkowo
  - Kamieniec Ząbkowicki
  - Lublin
- Puerto Rico (3):
  - Carolina
  - Rio Piedras
  - Río Grande
- Russia (6):
  - Kemerovo
  - Moscow
  - Ryazan
  - Saratov
  - Smolensk
  - Tyumen
- Spain (3):
  - Barcelona
  - Lleida
  - Oviedo
- United Kingdom (5):
  - Bath
  - Birmingham
  - Glasgow
  - Midsomer Norton
  - Rotherham